CLINICAL TRIAL: NCT02520622
Title: Evaluation of the Impact of Using Digital Photographs on a Mobile Device Versus Printed Photographs on Patient Conducted Skin Exams
Brief Title: Digital vs. Printed Photographs: Impact on Skin Self-Examinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 821426
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Experimental): Patients use digital photographs loaded onto a mobile device
  Interventions: Behavioral: Digital photographs loaded onto a mobile device
- Reminders (Experimental): Patients use digital photographs loaded onto a mobile device and receive skin exam reminders
  Interventions: Behavioral: Digital photographs loaded onto a mobile device; Behavioral: Skin exam reminders
- Social Support (Experimental): Patients use digital photographs loaded onto a mobile device and a social support network
  Interventions: Behavioral: Digital photographs loaded onto a mobile device; Behavioral: Social support network
- Combined (Experimental): Patients use digital photographs loaded onto a mobile device and a social support network and receive skin exam reminders
  Interventions: Behavioral: Digital photographs loaded onto a mobile device; Behavioral: Skin exam reminders; Behavioral: Social support network

INTERVENTIONS:
Behavioral: Digital photographs loaded onto a mobile device
Behavioral: Skin exam reminders
  Arms: Combined; Reminders
Behavioral: Social support network
  Arms: Combined; Social Support

SUMMARY:
The primary aim is to determine the impact of using digital photographs on a mobile device versus printed photographs on skin self-examination rates. The ease-of-use and overall satisfaction with the two exam modalities will be evaluated. Secondarily, the impact on melanoma thickness at detection, melanoma detection, biopsy, and office visit rates will be evaluated. The study involves patients in the Pigmented Lesion Clinic that have received total body photography for skin monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Penn Dermatology Pigmented Lesion Clinic who have a mobile device for personal use that either:
* (1) already have total body photography images, have a compact disc (CD) of digital versions of these images, and who do NOT already conduct proper monthly skin exams at home, and
* (2) patients that are having new images taken

Exclusion Criteria:

* Patients that are children or adolescents
* Patients that are court-ordered to attend residential alcohol or other drug treatment facilities and therefore considered prisoners
* Patients that are incompetent to provide informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Skin self-examination rates | 6 months
  Evaluate if printed photographs alone versus skin self-examinations supplemented with digital photos on a mobile device, or digital photos with reminders, social support networks, or both, lead to improved self-examination rates. This outcome is assessed by survey, before and after the intervention.

SECONDARY OUTCOMES:
Features important to a skin self-examination tool | 6 months
  Identify the features of digital or printed photograph use that are important to patients to have as part of a successful adjunct skin self-examination tool. This outcome is measured via survey after the intervention where participants rank on a Likert scale a series of features from critical to not important.
Melanoma thickness at detection | 6 months
  Determine if using printed photographs alone versus skin self-examinations supplemented with digital photos on a mobile device leads to differing melanoma thickness upon detection. This outcome will be assessed at the group level using descriptive statistics to calculate a mean thickness between the two groups where a Student's t-test will be used to assess significance.
Office visit rates | 6 months
  Determine if using printed photographs alone versus skin self-examinations supplemented with digital photos on a mobile device leads to differing office visit rates. This outcome will be assessed at the group level where the number of office visits over the course of the study will be compared for each group using a proportion's test or a chi-squared association test to assess if the rates between the two groups differ significantly.
Biopsy rates | 6 months
  Determine if using printed photographs alone versus skin self-examinations supplemented with digital photos on a mobile device leads to differing biopsy rates. This outcome will be assessed at the group level where the number of biopsies over the course of the study will be compared for each group using a proportion's test or a chi-squared association test to assess if the rates between the two groups differ significantly.
Melanoma detection rates | 6 months
  Determine if using printed photographs alone versus skin self-examinations supplemented with digital photos on a mobile device leads to differing melanoma detection rates. This outcome will be assessed at the group level where the number of new melanomas detected over the course of the study will be compared for each group using a proportion's test or a chi-squared association test to assess if the rates between the two groups differ significantly.
Study/technology implementation | 6 months
  Evaluate the study/technology implementation process using the implementation sciences RE-AIM framework to categorize and describe as follows:
  Reach
  1. Number of skin exams
  2. Number of first time skin exams
  3. Percent of patients offered/recommended full body photography
  Effectiveness a. (Please see the primary outcome variables)
  Adoption
  a. Percent opting for total body photography of whom it is offered/recommended
  Implementation
  1. Number and extent of changes to patient surveys
  2. Number and extent of changes to educational/training materials
  3. Number and percent of patients expressing interest in, or inquiring about the study
  4. Time spent educating patients on how to conduct a skin self-examination
  5. Time spent educating clinicians on the study
  Maintenance
  1. Number and percent of repeat skin exams
  2. Number and percent of patients abandoning a particular modality
  3. Changes in RE-AIM measurements from one month to the next

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Marek AJ, Chu EY, Ming ME, Khan ZA, Kovarik CL. Piloting the Use of Smartphones, Reminders, and Accountability Partners to Promote Skin Self-Examinations in Patients with Total Body Photography: A Randomized Controlled Trial. Am J Clin Dermatol. 2018 Oct;19(5):779-785. doi: 10.1007/s40257-018-0372-7. PMID 30062632